CLINICAL TRIAL: NCT03789617
Title: A Multi-center, Single-arm, Open, Phase I/IIa Clinical Trial to Evaluate the Efficacy and Safety of EBViNT Cell (EBV Specific Autologous CD8+ T Cell) in Patients With Treatment Failed Epstein Barr Virus (EBV)-Positive Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eutilex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EBViNT
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-04

CONDITIONS: EBV Associated Extranodal NK/T-cell Lymphoma; EBV-Associated GastricCarcinoma or Esophageal AdenoCarcinoma
Keywords: Cytotoxic T cell; Lymphoma; Immuno-oncology; ENKL; EBViNT; Gastric cancer; solid tumor; Esophageal AdenoCarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Lymphoma; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBViNT Cell (Experimental)
  Interventions: Biological: EBViNT Cell

INTERVENTIONS:
Biological: EBViNT Cell — 1. Dosage: 1 bag containing 1.4x10^9 cells/100mL
  2. Administration: Inject intravenously over 30 minutes
  3. Dosing schedule: Single dose
  Other Names: Eutil autologous blood-derived T lymphocytes

SUMMARY:
The present study is a multi-center, single-arm, open, phase I/IIa clinical trial to evaluate the efficacy and safety of EBViNT Cell when administered to patients with Epstein-Barr (EBV) positive malignancies The present study investigates with 5 parts; Part1-phase I: IP single therapy on ENKL and solid tumors Part2-phase I: IP + lymphodepletion on solid tumors Part 3&5- Phase IIa: IP single therapy on each ENKL and solid tumors Part 4- Phase IIa: IP + lymphodepletion on solid tumors

DETAILED DESCRIPTION:
The present study is a multi-center, single-arm, open, phase I/IIa clinical trial to evaluate the efficacy and safety of EBViNT Cell when administered to patients with Epstein-Barr (EBV) positive tumors

After proving the safety through Part 1 and part 2, the efficacy and safety would be studied through part 3~5.

* If CTCAE grade 3 or higher adverse drug events (ADR) do not occur in the three subjects: Begin enrollment for phase IIa
* If a CTCAE grade 3 or higher ADR occurs in one of the three subjects: Enroll three more subjects (up to six subjects in total) and assess whether any CTCAE grade 3 or higher ADR occurs

  * If a CTCAE grade 3 or higher ADR does not occur in the three additional subjects (1/6): Begin enrollment for phase IIa
  * If a CTCAE grade 3 or higher ADR occurs in at least one of the three additional subjects (more than 2/6): Begin enrollment for phase IIa at 7.0x10^8 cells, the maximum dose from phase I
* If a CTCAE grade 3 or higher ADR occurs in two of the three subjects: Begin enrollment for phase IIa at 7.0x10^8 cells, the maximum dose from phase I

Subjects participating in the present study will undergo 1) an EBV epitope screening test followed by 2) an eligibility assessment for clinical trial enrollment.

Subjects who are administered with the investigational product will be monitored until progressive disease (PD) is confirmed or for 24 weeks (main observation period of 4 weeks + monitoring for 20 weeks) to evaluate the product's safety and efficacy, and will undergo immunological assessment.

Radiological tests for tumor assessment will be conducted at the enrollment visit, 4 weeks, 8 weeks, 16 weeks, and 24 weeks and assessed by the Independent Radiology Review Committee (IRRC) using the Lugano criteria. To eliminate pseudo-progression, progressive disease (PD) will be determined by considering immunological tests, a quantitative EBV DNA assay, and intermediate response (IR) under LYRIC. Biopsies may be performed to achieve this.

ELIGIBILITY:
Inclusion Criteria (Visit 1)

1. At least 19 years of age
2. Patients with lymphomas or solid tumors who have been found to be positive for EBV encoded RNA (EBER) by in situ hybridization (ISH) (previous test results may be used as evidence if available)

   1. Part 1: Histologically or cytologically confirmed lymphoma or solid tumor
   2. Part 2: Histologically or cytologically confirmed solid tumor
   3. Part 3: Patients who have been diagnosed with histologically confirmed extranodal NK/T-cell lymphoma (ENKL) according to WHO classification
   4. Parts 4 and 5: Patients with histologically confirmed gastric cancer or esophageal adenocarcinoma
3. Patients who have given written consent to voluntarily participate in the epitope screening

Exclusion Criteria (Visit 1)

1. Patients with aggressive NK cell leukemia
2. Patients with hemophagocytic lymphohistiocytosis (HLH)
3. Persons who have previously received a solid organ transplant
4. Persons who have been diagnosed with a malignant tumor other than the target disease in the past 5 years (treated basal cell carcinoma, squamous epithelial cell carcinoma, and non-invasive cervical cancer do not necessitate exclusion)
5. Patients in whom a tuberculosis infection was confirmed in the 1 year prior to screening for the present study (However, patients who have been determined to be cured after treatment may be enrolled.)
6. Patients who test positive for anti-HIV antibodies
7. Patients deemed unsuitable to participate in the clinical trial by an investigator based on active infection (HBV, HCV) test results

Enrollment Criteria (Visit 2)

1. Persons who have been found to be capable of production in the epitope screening test
2. Patients who have failed standard treatment or conventional chemotherapy and who meet any one of the following

   1. Patients who have relapsed/progressed after 1 or more chemotherapies, and for whom standard treatment does not exist or cannot be performed
   2. Intolerable patients for whom anticancer treatment cannot be performed or a minimum of one full cycle cannot be completed in a first-line chemotherapy
   3. Patients who are refractory to first-line chemotherapy
3. Persons with evaluable lesions

   1. Lymphoma: Persons with at least 1 lesion with long axis > 15 mm or 18FDG-PET-CT avid
   2. Solid tumor: Persons with at least 1 measurable lesion based on RECIST 1.1
4. Persons with appropriate liver, renal, and bone marrow function (two retests are permitted for borderline results, and corrections such as transfusion are permitted)

Exclusion criteria (Visit 2)

1. Where central nervous system (CNS) lymphoma or uncontrolled CNS metastasis is present (patients with brain metastasis that has been treated and is stable [stable for at least 30 days based on radiology records] may be enrolled)
2. Persons who have received surgery, radiotherapy, or chemotherapy in the 3 weeks prior to the investigational product administration
3. Persons who have been administered any other investigational product in the 3 weeks prior to the investigational product administration
4. Persons who have not recovered from the toxicity of any previous treatment to Grade 1 or lower based on NCI CTCAE v5.0 (however, clinically insignificant toxicities such as alopecia are excluded)
5. Patients who have received immunosuppressants, including steroids, in the 10 days prior to blood collection (Visit 2) for production of the study drug (however, local steroids and steroids for inhalers are permitted, and steroid equivalent to 20 mg/day of prednisolone may be administered at the investigator's discretion)
6. Patients with the following (but not limited to) clinically significant cardiovascular comorbidities as determined by the investigator

   : Uncontrolled hypertension (i.e., systolic pressure > 180 mmHg and/or diastolic pressure > 100 mm/Hg), unstable angina, pulmonary embolism, cerebrovascular disease, valvular disease, congestive heart failure (NYHA severity classification Grade III or IV), or myocardial infarction or serious cardiac arrhythmia within the 24 weeks prior to the enrollment visit
7. Patients with findings of autoimmune or inflammatory disease, whose abnormal results from an autoimmune response test have been deemed clinically significant by an investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Confirmed objective response rate (confirmed ORR) [assessed by IRRC] | up to 6 month from LPI

SECONDARY OUTCOMES:
Duration of response (DoR) [assessed by IRRC and investigator] | up to 6 month from LPI
Disease control rate (DCR) [assessed by IRRC and investigator] | up to 6 month from LPI
Objective response rate (ORR) [assessed by investigator] | up to 6 month from LPI
Complete response rate (CR rate) [assessed by IRRC and investigator] | up to 6 month from LPI
Partial response rate (PR rate) [assessed by IRRC and investigator] | up to 6 month from LPI
Partial response duration (PR duration) [assessed by IRRC and investigator] | up to 6 month from LPI
Progression-free survival (PFS) | up to 6 month from LPI
Overall survival (OS) | up to 6 month from LPI

OTHER OUTCOMES:
Immunological assessment | up to 6 month
  Plasma cytokine analysis (IL-1b, IL-2, IL-4, IL-6, IL-8, IL-10, TNF, IFN-γ, IL-17a) EBV LMP2a-specific cytokine production (IL-1b, IL-2, IL-4, IL-6, IL-8, IL-10, TNF, IFN-γ, IL-17a) Phenotypical analysis of CD8 T cells
Quantitative EBV DNA assay | up to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Seok Eom, MD, Principal Investigator — National Cancer Center; Won Seog Kim, MD, Principal Investigator — Samsung Medical Center; Ho Jin Shin, MD, Principal Investigator — Pusan National University Hospital; Min-hee Ryu, MD, Principal Investigator — Asan Medical Cente; Won Sik Lee, MD, Principal Investigator — Inje University; Minsuk Kwon, MD, Principal Investigator — Ajou Univ. Hosp.; Hyo song Kim, MD, Principal Investigator — Severance Hosp; Jeeyun Lee, MD, Principal Investigator — Samsung Medical Center
Locations (8):
- South Korea (8):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Inje Univ. Hosp, Pusan
  - Pusan national Univ. Hosp., Pusan
  - Samsung Medical Center, Seoul
  - Seoul Asan Medical center, Seoul
  - Severance hosp., Seoul
  - Ajou Univ Hosp., Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eom HS, Choi BK, Lee Y, Lee H, Yun T, Kim YH, Lee JJ, Kwon BS. Phase I Clinical Trial of 4-1BB-based Adoptive T-Cell Therapy for Epstein-Barr Virus (EBV)-positive Tumors. J Immunother. 2016 Apr;39(3):140-8. doi: 10.1097/CJI.0000000000000113. PMID 26938947
- [Background] Choi BK, Lee SC, Lee MJ, Kim YH, Kim YW, Ryu KW, Lee JH, Shin SM, Lee SH, Suzuki S, Oh HS, Kim CH, Lee DG, Hwang SH, Yu EM, Lee IO, Kwon BS. 4-1BB-based isolation and expansion of CD8+ T cells specific for self-tumor and non-self-tumor antigens for adoptive T-cell therapy. J Immunother. 2014 May;37(4):225-36. doi: 10.1097/CJI.0000000000000027. PMID 24714356
- See also: Web address — http://www.eutilex.com/en/